CLINICAL TRIAL: NCT00096876
Title: Screening Evaluations for Neurologic Syndromes: Olfactory Testing in Relatives of Parkinson's Disease Patients
Brief Title: A Study of the Sense of Smell in Relatives of Parkinson's Disease Patients
Status: Completed | Type: Observational
Sponsor: Institute for Neurodegenerative Disorders (Other)
Responsible Party: Sponsor
Other Study IDs: SENSOR
Record Dates: First submitted 2004-11-16; First posted 2004-11-17 (Estimated); Last update posted 2019-04-03 (Actual); Status verified 2019-04

CONDITIONS: Parkinson Disease; Parkinsonian Syndrome
Keywords: Parkinsonian syndrome
MeSH Terms: conditions — Parkinson Disease; Parkinsonian Disorders

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
In this study, individuals complete and return a mail survey, specifically a 40 item scratch and sniff smell test.

DETAILED DESCRIPTION:
This study would extend the findings of previous studies by characterizing the performance of the 40-item UPSIT in a cohort of first-degree relatives of Parkinson's disease (PD) patients. The results would also validate the use of the University of Pennsylvania Smell Identification Test (UPSIT) as a mail-survey instrument. Once identified, these individuals could be followed as a potentially at-risk cohort to determine if the screening evaluation was predictive of later developing Parkinson's disease. The results from this pilot study have the potential to guide the use of olfactory testing using the UPSIT as a screening tool, and to provide necessary preliminary data for planning clinical trials to prevent the occurrence of PD in at-risk individuals.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be a first-degree relative of a PD patient with diagnosis confirmed by a movement disorders specialist at the Institute for Neurodegenerative Disorders
* Subject must not carry a diagnosis of PD or other neurodegenerative disorder
* Subject must be either at least 50 years old or within 10 years of the age of onset of their affected relative
* Subject must be a non-smoker
* Subject must have no other known reason for abnormal olfaction (e.g. nasal trauma)

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2004-10; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Danna Jennings, MD, Principal Investigator — Institute for Neurodegenerative Disorders
Locations (1):
- Institute for Neurodegenerative Disorders, New Haven, Connecticut, United States

REFERENCES:
- [Background] Berendse HW, Booij J, Francot CM, Bergmans PL, Hijman R, Stoof JC, Wolters EC. Subclinical dopaminergic dysfunction in asymptomatic Parkinson's disease patients' relatives with a decreased sense of smell. Ann Neurol. 2001 Jul;50(1):34-41. doi: 10.1002/ana.1049. PMID 11456307
- [Background] DeKosky ST, Marek K. Looking backward to move forward: early detection of neurodegenerative disorders. Science. 2003 Oct 31;302(5646):830-4. doi: 10.1126/science.1090349. PMID 14593169
- [Background] Doty RL, Shaman P, Dann M. Development of the University of Pennsylvania Smell Identification Test: a standardized microencapsulated test of olfactory function. Physiol Behav. 1984 Mar;32(3):489-502. doi: 10.1016/0031-9384(84)90269-5. PMID 6463130
- [Background] Doty RL, Bromley SM, Stern MB. Olfactory testing as an aid in the diagnosis of Parkinson's disease: development of optimal discrimination criteria. Neurodegeneration. 1995 Mar;4(1):93-7. doi: 10.1006/neur.1995.0011. PMID 7600189
- [Background] Marek KL, Seibyl JP, Zoghbi SS, Zea-Ponce Y, Baldwin RM, Fussell B, Charney DS, van Dyck C, Hoffer PB, Innis RP. [123I] beta-CIT/SPECT imaging demonstrates bilateral loss of dopamine transporters in hemi-Parkinson's disease. Neurology. 1996 Jan;46(1):231-7. doi: 10.1212/wnl.46.1.231. PMID 8559382
- [Background] Markopoulou K, Larsen KW, Wszolek EK, Denson MA, Lang AE, Pfeiffer RF, Wszolek ZK. Olfactory dysfunction in familial parkinsonism. Neurology. 1997 Nov;49(5):1262-7. doi: 10.1212/wnl.49.5.1262. PMID 9371905
- [Background] Montgomery EB Jr, Baker KB, Lyons K, Koller WC. Abnormal performance on the PD test battery by asymptomatic first-degree relatives. Neurology. 1999 Mar 10;52(4):757-62. doi: 10.1212/wnl.52.4.757. PMID 10078723
- [Background] Morrish PK, Rakshi JS, Bailey DL, Sawle GV, Brooks DJ. Measuring the rate of progression and estimating the preclinical period of Parkinson's disease with [18F]dopa PET. J Neurol Neurosurg Psychiatry. 1998 Mar;64(3):314-9. doi: 10.1136/jnnp.64.3.314. PMID 9527140
- [Background] Mouradian MM. Recent advances in the genetics and pathogenesis of Parkinson disease. Neurology. 2002 Jan 22;58(2):179-85. doi: 10.1212/wnl.58.2.179. PMID 11805242
- [Background] Quinn NP, Rossor MN, Marsden CD. Olfactory threshold in Parkinson's disease. J Neurol Neurosurg Psychiatry. 1987 Jan;50(1):88-9. doi: 10.1136/jnnp.50.1.88. PMID 3819760